CLINICAL TRIAL: NCT04520477
Title: Watershift - Pilot Study: Observing the Interindividual Effects and Mechanims of the Uptake, Storage and Excretion of Water
Brief Title: Watershift - Pilot Study
Acronym: WATERSHIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EC2017/1636
Record Dates: First submitted 2020-08-11; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Total Body Water; Nocturnal Polyuria
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bio Impedance assesement (BIA) — BIA every 5 minutes od the test protocol. Patients stood up for 5 minutes, laid down for 70 minutes, followed by 5 minutes in a seated position and ending with 30 minutes standing. BIA was done every 5 minutes.
Diagnostic Test: Blood and salava sample — Blood Samples were done at the initation of the protocol, and every 10 minutes after ingestion of the deutarated water
Dietary Supplement: Ingestion of deuterated water — 15 minutes after the intiation of the test protocol, participants drink an amount of deuterated water corresponding with 0.25% of their TBW calculated using the Watson Formula
Diagnostic Test: Urine sample — A urine sample is taken at the initiation and after termination of the protocol.

SUMMARY:
The aim of this pilot was to study how body water behaves between the different internal water pools of the human body, what the role and influence of the interstitium is and what the effect is of body position on the distribution and allocation of BW between different body parts (trunk, legs, arms). To study this, 2 techniques that have not been used before in urological research were tested on their usefulness:

* The first technique is a recent BIA device, which distinguishes itself from earlier devices by measuring impedance at different electrical currencies in different body parts (arm/limb/trunk). This technique made it possible to observe the influence of body position on the distribution of BW in these body compartments. Rationale for this research question is mainly the link between NP and edema that was found in earlier research and the fact that body position seemed to have an impact on the size of edema. For this reason, it can be suggested that body position and thus edema will have an impact on whether or not NP occurs.
* The second technique uses deuterium as a biological marker. With this technique the distribution, storage, allocation and excretion of BW was examined among the urological most relevant water pools (blood, urine and interstitium).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Ages between 18 and 30
* BMI between 18 and 24.9

Exclusion Criteria:

* Intake of medications except of OAC
* Patients with pacemaker or neurostimulator

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Observing the absorption time, and the lay over time from deuterated water from the gast of deuterated water in the blood | 3 hours
  Aim of this overview is to assess how fast the deuterium oxide ingested in the human gastro-intestinal tractus, the colon and the blood pool. We want to know if this is 5min or even more 30 min and when the maximal dose of deuterium in the blood is reached.
Observing impedance changes linked with position switch | 5 minutes
  Decrease of impedance by 1 amplitude by changing positions grom standing to lying.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided